CLINICAL TRIAL: NCT03769870
Title: A Randomized, Open-label, Cross-over, Multiple Dosing Study to Evaluate Drug-drug Interaction Between Teneligliptin and Atorvastatin in Healthy Male Adults
Brief Title: Teneligliptin and Atorvastatin DDI Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MP_C104
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teneligliptin (Other)
  Interventions: Drug: Teneligliptin 20mg/day
- Atorvastatin (Other)
  Interventions: Drug: Atorvastatin 40mg/Day
- Teneligliptin + Atorvastatin (Other)
  Interventions: Drug: Teneligliptin 20mg/day + Atorvastatin 40mg/day

INTERVENTIONS:
Drug: Teneligliptin 20mg/day — cross-over
  Arms: Teneligliptin
Drug: Atorvastatin 40mg/Day — cross-over
  Arms: Atorvastatin
Drug: Teneligliptin 20mg/day + Atorvastatin 40mg/day — cross-over
  Arms: Teneligliptin + Atorvastatin

SUMMARY:
A randomized, open-label, cross-over, multiple dosing study to evaluate drug-drug interaction between Teneligliptin and Atorvastatin in healthy male adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adult 19 to 45 years
2. Body weight ≥ 50kg, and BMI between 18-29kg/m2 at screening
3. Subject who agrees to use a medically acceptable double-barrier method of contraception and not to donate sperms from the first dose until 2 months after the last dose.
4. Subject who was given, and fully understood, the information about the study, and has provided voluntary written informed consent to participate in the study and agreed to comply with the study requirements.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Cmax,ss(Maximum concentration at steady state) | 24 hours
AUCτ,ss(Area under the concentration-time curve at steady state) | 24hours

CONTACTS AND LOCATIONS:
Locations (1):
- Korea Universitiy Guro Hospital, Seoul, South Korea